CLINICAL TRIAL: NCT06901713
Title: Protocol for a Smoking Cessation Program With CBT Text and Mindfulness Audio Support: A Randomized Controlled Trial
Brief Title: Smoking Cessation Program With CBT and Mindfulness Audio Support: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-2068-01
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-02

CONDITIONS: Smoking Cessation; Tobacco Dependence
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT text-based program alone (Active Comparator): Participants in this group will receive CBT text messages focused on smoking cessation strategies, including identifying triggers, developing coping mechanisms, and setting goals. These messages will be sent at regular intervals over the course of the 8-week program.
  Interventions: Other: cognitive behaviour thearpy
- CBT text combined with mindfulness audio (Experimental): In addition to the CBT text messages similar to Group A, participants in this group will also have access to a series of mindfulness audio recordings. These recordings will guide participants through mindfulness exercises such as body scans, breath awareness, and meditation, designed to enhance self-awareness and emotion regulation in the context of smoking cessation. The audio will be provided weekly, corresponding to the weekly themes of the program. Participants in this group will receive emotional support and peer-related information from chatbots.
  Interventions: Other: cognitive behaviour thearpy; Other: mindfulness

INTERVENTIONS:
Other: cognitive behaviour thearpy — Participants will access the CBT text materials through a dedicated platform
Other: mindfulness — Participants will access the mindfulness audio via a compatible device
  Arms: CBT text combined with mindfulness audio

SUMMARY:
This protocol describes a randomized controlled trial evaluating the effectiveness of a smoking cessation program with two intervention methods. One method provides only CBT text messages (Group A), while the other combines CBT text with mindfulness audio (Group B). The study aims to compare the two approaches in reducing smoking frequency, managing cravings, and improving emotional regulation.

This study investigates the effects of two different smoking cessation interventions: (1) CBT text-based program alone (Group A), and (2) CBT text combined with mindfulness audio (Group B). The primary outcomes include reductions in smoking frequency and cravings, as well as improvements in emotional regulation and quality of life.

DETAILED DESCRIPTION:
Design: A randomized controlled trial (RCT) will be used to compare the outcomes of the two intervention groups.

Setting: The study will be conducted online. Participants will access the CBT text materials through a dedicated platform and the mindfulness audio via a compatible device. Recruitment will be done through social media, community outreach, and online advertisements.

ELIGIBILITY:
Inclusion Criteria:

* Who smoke at least 5 cigarettes per day.
* Express a desire to quit or reduce smoking.
* Who has the ability to access and use the provided digital materials.

Exclusion Criteria:

* Those currently enrolled in other smoking cessation programs.
* Individuals with severe psychiatric disorders that may interfere with participation.
* Those without access to the necessary digital devices.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Biological Verification of Abstinence | 6 Months
  Confirmation of smoking abstinence at the end of the study period using cotinine test strips. This will be the main measure to assess the effectiveness of the smoking cessation interventions.

SECONDARY OUTCOMES:
Smoking Frequency | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 26.
  Measured by the number of cigarettes smoked per day at baseline
Craving Intensity | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 26.
  Assessed using a visual analog scale (VAS)
Emotional Regulation | Baseline, Week 12, and Week 26
  Evaluated using the Depression, Anxiety, and Stress Scale (DASS-21)

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li S, Meng L, Chiolero A, Ma C, Xi B. Trends in smoking prevalence and attributable mortality in China, 1991-2011. Prev Med. 2016 Dec;93:82-87. doi: 10.1016/j.ypmed.2016.09.027. Epub 2016 Sep 24. PMID 27677441
- [Background] Li Q, Hsia J, Yang G. Prevalence of smoking in China in 2010. N Engl J Med. 2011 Jun 23;364(25):2469-70. doi: 10.1056/NEJMc1102459. No abstract available. PMID 21696322